CLINICAL TRIAL: NCT06579859
Title: PNRR-MR1-2023-12377031, Development of a Registry to Assess Natural History in Duchenne Muscular Dystrophy
Brief Title: Development of a Registry to Assess Natural History in Duchenne Muscular Dystrophy
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6906
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: None Retained — dna
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Duchenne muscular dystrophy is a rare progressive X-linked neuromuscular disease, caused by mutation in the dystrophin gene, leading to progressive muscle degeneration, loss of specific functional milestones, severe respiratory and cardiac impairment. Improved standards of care and the regular early use of glucocorticoid treatment have changed the natural history of the disease, affecting both survival and the time of loss of functional milestones. More recently, there has been increasing evidence of an additional benefit from new therapeutical approaches based on mechanisms targeting specific type of mutation; therefore, it has become mandatory to obtain more detailed long-term information about the patterns of progression related to different genotypes. The aim of this project is to better define the natural history of Duchenne musculare Dystrophy patients and to understand clinical and motor functional trajectories defining a more specific genotype/phenotype characterization according to the type of mutation.

DETAILED DESCRIPTION:
Duchenne muscular Dystrophy is a progressive disorder affecting one in 3600-5000 live male births, leading to a progressive loss of specific functional milestones.

Over the past two decades, the development of new outcome measures has allowed a better definition of the natural history of the disease. Recently, there has been increasing evidence of benefit from new therapeutical approaches based on inflammatory, fibrotic and genetic mechanisms targeting specific type of mutations. The changes are better observed after the first year of treatment but as it is not possible to maintain placebo for such a long time, it has become mandatory to have natural history data for comparison. As there is increasing evidence that specific groups of mutations may have different progression of the disease, a few studies have been performed to study longitudinal functional changes in Duchenne patients with different types of mutations (deletion, duplication, small mutations) and in the subgroups eligible for skipping individual exons, focusing on those skipping 44, 45, 51 and 53 . Our groups has been involved in national and international efforts to define the trajectories of progression according to phenotypes, reporting functional changes using different measures such as the six minute walking test , North Star Ambulant Assessment in ambulant patients, and in non-ambulant patients, using the Performance of Upper limb test 2.0 and respiratory function.

The study will involve all patients with genetically confirmed Duchenne muscular Dystrophy diagnosis currently in follow up in 4 italian centers.

This research aims to provide more information about natural history in Duchenne patients, including genetic, functional motor, cardiological and respiratory data collection to define a better and complete genotype and phenotype correlation, not only in ambulant but also in not ambulant patients.

ELIGIBILITY:
Inclusion Criteria:

* patient with genetic confirmation od Duchenne Muscular Dystrophy in follow up in one of the 4 involved centers
* signed informed consent form

Exclusion Criteria:

* patients who refuses consent

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: males affected by Duchenne Muscular Dystrophy in regular already in follow up or enrolled in one of the four involved center for neuromuscular disorders who will attend regular follow up visits as for standard of care will be enrolled in the study
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
integrate existing datasets | 3 years
  To integrate the existing datasets including 3 year follow up data of ambulant Duchenne patients with new patients having at least 3 year follow up and with further follow up achieved after the study was completed. The dataset will also include data on non ambulant patients
Develop structurate Case Report Form | 3 years
  To develop a structured electronic Case Report Form that will include all the functional data such as 6 Minute Walking Test ( no scaled) , North Star Ambulatory Assesment ( scale 0-34), timed items ( not scaled) , Performance Upper Limb (0-42) collected as part of the clinical routine and other clinical and genetic variables routinely collected and available from clinical notes.
  To transfer the existing data to the newly developed Case report form
analyse clinical data | 3 years
  To analyse 3 years data follow up in the original cohort and in all those who have more than 3 year follow up
  In patients who lost ambulation during the study, their retrospective functional data will be analysed looking for possible prognostic indicators at one, two and three years before loss of ambulation

CONTACTS AND LOCATIONS:
Overall Officials: Marika Pane, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (4):
- Italy (4):
  - ASL LANCIANO VASTO CHIETI, Laboratorio di Patologie Neuromuscolari del Centro di Riferimento Regionale per le Malattie Neuromuscolari, Chieti, Ch
  - ASST Grande Ospedale Metropolitano Niguarda, Centro Clinico Nemo Milano, Milan, MI
  - Azienda Ospedaliera Universitaria "G. Martino"UOC di Neurologia e Malattie Neuromuscolari, Messina
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC NEMO Pediatrico, Roma